CLINICAL TRIAL: NCT07046572
Title: A Double-blind Placebo-controlled Randomized Controlled Trial (RCT) of 3ml Methoxyflurane for Intrauterine Device (IUD) Insertion and Endometrial Biopsy
Brief Title: Methoxyflurane for IUD Insertion and Endometrial Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Matthew Morton Research Award (Unknown)
Responsible Party: Principal Investigator, Mara Sobel, Principal Investigator (Dr.), Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: REB 25-0041-A
Record Dates: First submitted 2025-06-20; First posted 2025-07-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Biopsy; Intrauterine Devices
Keywords: methoxyflurane

STUDY DESIGN:
Intervention Model Description: The proposed study is a double-blind randomized controlled trial. Participants will be recruited from Mount Sinai Hospital outpatient gynecology clinics. Recruitment, consent, randomization, procedure, and post-procedure survey will occur during the same visit. Each participant will be randomly assigned to one of two arms: 1) intervention (3ml of Methoxyflurane via a Penthrox inhaler) or 2) placebo (3ml of normal saline via an identical placebo Penthrox inhaler). The primary outcome will be a global pain score, which will be patient-reported by the 100 mm Visual Analogue Scale (VAS) following the procedure.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The research coordinator (who is not involved in direct patient care) will open the allocation envelopes without the presence of the participant or the provider. They will prepare the Penthrox inhalers with either 3 mL methoxyflurane or 3 mL normal saline with a few drops of methoxyflurane on the outside of the inhaler to maintain blinding (as methoxyflurane has a distinct smell). The research coordinator will label each Penthrox inhaler with the study ID number.
  The provider (who is blinded to the study) will enter the patient room with the procedure tray and the Penthrox inhaler. They will instruct the patient to inhale for 10 breaths with their finger covering the dilutor hole of the Penthrox inhaler. Once the patient has taken 10 breaths, the research assistant will start a timer for 5 minutes. The research assistant will inform the OB-GYN once the 5 minutes have passed and at that point the OB-GYN will start the procedure. All data will remain blinded until data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3ml of Methoxyflurane (Experimental): 3ml of Methoxyflurane via a Penthrox inhaler
  Interventions: Drug: Methoxyflurane - Penthrox
- 3ml of normal saline (Placebo Comparator): 3ml of normal saline via an identical placebo Penthrox inhaler
  Interventions: Other: Placebo Penthrox inhaler

INTERVENTIONS:
Drug: Methoxyflurane - Penthrox — 3ml of Methoxyflurane via a Penthrox inhaler
  Arms: 3ml of Methoxyflurane
Other: Placebo Penthrox inhaler — 3ml of normal saline via an identical placebo Penthrox inhaler
  Arms: 3ml of normal saline

SUMMARY:
The aim of this study is to determine if 3ml of inhaled Methoxyflurane, in the form of a Penthrox inhaler, reduces pain during IUD insertion and/or endometrial biopsy. The proposed study is a double-blind, placebo-controlled RCT.

Each participant will be randomly assigned to one of two arms:

1. Intervention (3ml of Methoxyflurane via a Penthrox inhaler)
2. Placebo (3ml of normal saline via an identical placebo Penthrox inhaler)

The primary outcome is global pain score, which will be patient-reported by the 100 mm Visual Analogue Scale (VAS) 5-minutes following the procedure (endometrial biopsy or IUD insertion).

ELIGIBILITY:
Inclusion Criteria

* Any participant ≥18 years and ≤ 65 years presenting for an IUD insertion or endometrial biopsy
* For IUD insertion, only nulliparous patients
* English speaking participants only
* Availability of a ride home from the appointment

Exclusion Criteria

* Use of pain medication that is not an NSAID or acetaminophen (e.g. opioids, benzodiazepines) within past 24 hours
* Misoprostol administration within 24 hours
* Breastfeeding
* Any diagnosed chronic pain syndromes (e.g. fibromyalgia, vaginismus)
* Allergy to methoxyflurane
* Renal or liver disease
* Known or genetically susceptible to malignant hyperthermia or a history of severe adverse reactions in either patient or relatives
* Baseline vital signs of systolic blood pressure <100, diastolic blood pressure <60 and/or pulse <60.
* Previous unsuccessful office attempt of IUD insertion or endometrial biopsy by the same practitioner (note of clarification: previous unsuccessful IUD insertion or biopsy attempt by a different practitioner will still be eligible)
* Clinically evident respiratory impairment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Global pain score | 5-minutes following the completion of the procedure
  Patient reported pain by the 100 mm Visual Analogue Scale (VAS), minimum value 0 (no pain at all) and maximum value 100 (worst pain imaginable), higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Pain scores during procedure | During the procedure
  Patient-reported verbal pain scores on a scale from 0 (no pain) to 10 (worst pain imaginable) at the following timepoints: baseline before inhaler, baseline after inhaler, insertion of speculum, tap cervix with sound, placement of tenaculum, sounding (IUD only), IUD insertion/endometrial biopsy, and 1-minute post-procedure. Higher scores indicate greater pain intensity.
Immediate complications and side effects | Immediately after the completion of the procedure
  Provider-reported via written survey
Difficulty for provider to complete the procedure | Immediately after the completion of the procedure
  Provider-reported on Likert scale, minimum 1 (least difficult) and maximum 5 (most difficult). Higher score indicates greater difficulty.
Length of time for procedure completion | During the procedure
  Recorded via stopwatch
Patient satisfaction | Immediately after the completion of the procedure
  Patient-reported via a written survey
Patient Satisfaction | Immediately after the completion of the procedure
  Patient-reported via a 5-point Likert scale: very unsatisfied (1) to very satisfied (5). Higher score indicates greater dissatisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- OPG, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No